CLINICAL TRIAL: NCT05325242
Title: Safety and Efficacy of Elbow Artery Embolization (EAE) for the Treatment of Lateral Epicondylitis
Brief Title: Elbow Artery Embolization for Tennis Elbow
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Siddharth Padia, MD (Other)
Responsible Party: Sponsor-Investigator, Siddharth Padia, MD, Professor of Radiology, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-000161
Record Dates: First submitted 2022-02-17; First posted 2022-04-13 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Lateral Epicondylitis, Unspecified Elbow
Keywords: tennis elbow; embolization; embozene
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Elbow Artery Embolization (EAE) (Experimental): Patients will undergo EAE with Embozene microspheres (75 micron). The microspheres will be delivered in a saline-contrast medium solution and will be delivered to the arteries supplying the areas of the patient's pain.
  Interventions: Device: Embozene particles

INTERVENTIONS:
Device: Embozene particles — Embozene particles are FDA approved for the embolization of hypervascular tumors and arteriovenous malformations. Several studies have shown excellent safety and efficacy with regards to tumor control and objective response in liver cancer. It has been used extensively for the treatment of symptomatic uterine fibroids, where Embozene embolization of the uterine arteries results in necrosis of uterine fibroids and cessation of abnormal vaginal bleeding. Other proven uses include embolization of arteriovenous malformations and fistulas.

SUMMARY:
The purpose of this clinical research study is to examine whether embolization treatment of an elbow artery is a safe and effective way to treat elbow pain, specifically pain from tennis elbow. Embozene is a medical device made by Varian marketed in the United States for the treatment of hypervascular tumors and arteriovenous malformations. It consists of thousands of microscopic spheres that are injected into the artery to block the flow of blood to a specific region. One of the causes of pain in the setting of tennis elbow is increased blood flow going to the specific area of pain. In this study, we will investigate an experimental procedure to decrease the blood flow (embolize) to the specific region of the elbow that is causing the pain. This will be done by infusing Embozene particles into the specific blood vessel supplying the area of pain in the elbow. This is an investigational study to evaluate the safety and efficacy of elbow artery embolization (EAE) for the treatment of symptomatic lateral epicondylitis (tennis elbow).

DETAILED DESCRIPTION:
This is a single-center, prospective, single arm investigational study to evaluate the safety of elbow artery embolization (EAE) for treatment of symptomatic lateral epicondylitis. In addition, the improvement as part of efficacy will be reported. All patients will have either failed or be intolerant to conservative management. Patients will be considered enrolled in the study once they have provided informed consent and have been determined to meet all eligibility criteria. A total of 25 patients will be enrolled in the single treatment arm of the study and will be followed for 24 months.

The study will involve a screening period in which patient eligibility is determined. Once eligibility is confirmed, subjects will undergo EAE with Embozene microspheres (75 micron). Following treatment, subjects will return for follow-up visits at 1 week, 1 month (± 2 weeks), 3 months (± 2 weeks), 6 months (± 4 weeks), 12 months (± 4 weeks), and 24 months (± 4 weeks) post-procedure. At these visits, subjects will undergo a directed physical examination, report any new adverse events (AEs), and complete questionnaires. At 12 months of follow-up, subjects will also undergo elbow MRI and x-ray.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of lateral epicondylitis based on history and physical exam
* Ability to provide informed consent
* Life expectancy greater than 12 months
* Moderate-severe lateral elbow pain as determined by visual analog scale > 4 (based on average severity during physical activity)
* Resistant/failed conservative treatment (e.g. NSAIDS/physical therapy/steroid joint injection) for at least 6 months.

Exclusion Criteria:

* Mild elbow pain as determined by visual analog scale < 4
* Chronic renal insufficiency (serum creatinine >2 mg/dL)
* Allergy to iodinated contrast agents that is not responsive to steroid management
* Active Infection or malignancy
* Prior elbow surgery in the subject elbow
* Uncorrectable bleeding diathesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Assess the efficacy of EAE in treating pain measured as percentage of subjects with a greater than 50% decrease in QuickDASH (Disabilities of the Arm, Shoulder, and Hand) score at 12 months. | 12 months
  Changes in QuickDASH (Disabilities of the Arm, Shoulder, and Hand) score as a measure of efficacy.

SECONDARY OUTCOMES:
Changes in Visual Analog Scan (VAS) as a measure of efficacy | 24 months
  The Faces Pain Scale is a numerical self-report measure of pain intensity developed for children to score the sensation of pain from 0-10. Pictures of 6 cartoon faces ranging from neutral expression of "no pain" (0) to "very much pain" (10). Participant is asked to point to the face that shows how much participant hurts at the time of assessment.
Change in symptoms as assessed by the QuickDASH scores. | 24 months
  the QuickDASH (Disabilities of the Arm, Shoulder, and Hand) uses 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb. each item has 5 response options, ranging from 1 (no difficulty) to 5 (unable) and, from the item scores, scale scores are calculated, ranging from 0 (no disability) to 100 (most severe disability)
Change in symptoms as assessed by the patient-rates tennis elbow evaluation (PRTEE) scores. | 24 months
  Patient-Rated Tennis Elbow Evaluation (PRTEE) is a 15-item questionnaire designed to measure forearm pain and disability in patients with lateral epicondylitis. The PRTEE allows patients to rate their levels of tennis elbow pain and disability from 0 to 10 ("0" being no pain, and "10" being worst imaginable).
Change in imaging | 12 months
  Change in radiographic imaging by elbow MRI and elbow radiograph

CONTACTS AND LOCATIONS:
Overall Officials: Siddharth Padia, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided